CLINICAL TRIAL: NCT01856088
Title: Stents Coated With the Biodegradable Polymer on Their Abluminal Faces and Elution of Sirolimus Versus Biolimus Elution for the Treatment of de Novo Coronary Lesions - Destiny Trial
Brief Title: DESTINY TRIAL (Inspiron x Biomatrix)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scitech 004
Record Dates: First submitted 2012-12-27; First posted 2013-05-17 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery; Drug eluting stent; thrombosis
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiron Stent (Experimental): Stent Inspiron with Sirolimus
  Interventions: Device: Inspiron Stent
- Biomatrix Flex Stent (Active Comparator): Stent Biomatrix Flex with biolimus
  Interventions: Device: Biomatrix Flex Stent

INTERVENTIONS:
Device: Inspiron Stent — stent implantation
  Other Names: Angioplasty
  Arms: Inspiron Stent
Device: Biomatrix Flex Stent — stent implantation
  Other Names: Angioplasty
  Arms: Biomatrix Flex Stent

SUMMARY:
The main objective of this study is to evaluate the effectiveness of stent Inspiron ™ sirolimus-eluting and coating the abluminal biodegradable stent Biomatrix Flex ™ lesions in native coronary arteries.

DETAILED DESCRIPTION:
This is a study of non-inferiority, multicentre, prospective, randomized into two treatment arms: I) Inspiron ™ stent eluting sirolimus or II) ™ Biomatrix stent eluting biolimus. Are a total of 165 randomized patients.

Patients will be followed for 60 months after the procedure. All new patients will be undergoing angiography for evaluation at 9 months. A subgroup of 60 patients will be evaluated with volumetric intravascular ultrasound at 9 months. Also, a subgroup of 21 patients will be evaluated with optical coherence tomography at the end of the index procedure and 9 months. It is anticipated that the total study duration is 72 months: 12 months to complete the admission of patients and 60 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Symptomatic ischemic heart disease and / or objective evidence of myocardial ischemia with one or two target lesions located in different epicardial vessels;
3. A(s) lesion(s) to target(m) must be:

   1. Again (not restenotic);
   2. Located in a native coronary artery diameter from 2.5 to 3.5 mm (visual);
   3. Can be treated with a single stent up to 29 mm in length;
   4. Obstruction with stenosis > 50% diameter (visual);
4. Acceptable candidate for CABG;
5. The patient will be informed of the nature of the study, agree with their rules and provide a written informed consent approved by the local Ethics Committee.

Exclusion Criteria:

1. Women of childbearing age with no history of surgical sterilization;
2. Myocardial infarction with Q wave occurred in the last 48 hours before the index procedure;
3. Myocardial infarction with or without Q wave with cardiac markers even at high levels;
4. Ejection fraction < 30%;
5. Impaired renal function (creatinine> 2.0 mg / dl) or calculated creatinine clearance < 60 ml / min;
6. Platelet count <100,000 cells/mm3 or > 700,000 cells/mm3;
7. Total leukocyte count <3000 cells/mm3;
8. Documented or suspected liver disease (including laboratory evidence of hepatitis);
9. Heart transplant recipient;
10. Known allergies to aspirin, clopidogrel, ticlopidine, paclitaxel, sirolimus, heparin or stainless steel;
11. Patient with a life expectancy less than 12 months;
12. Any significant medical condition which in the opinion of the investigator would interfere with the ideal of patient participation in this study;
13. Participation in other research in the last 12 months, unless there is direct benefit to the research subject;
14. Coronary angioplasty (with or without stenting) for less than 6 months anywhere in the target vessel;
15. Coronary angioplasty (with or without stenting) prior to any time in that segment Diste less than 5 mm (proximal or distal) of the lesion;
16. Coronary angioplasty (with or without stenting) scheduled in the first 12 months after the index procedure in any segment of the target vessel.

EXCLUSION CRITERIA angiographic

1. Restenotic target lesion;
2. Need for treatment for more than one lesion in the same vessel;
3. Need for treatment with three or more lesions in the same procedure;
4. Target vessel diameter <2.5 mm or> 3.5 mm (visual);
5. Target lesion long not susceptible to treatment with a single stent to 29mm in length, according to the judgment of the operator;
6. Lesion of the coronary artery unprotected ( > 50% stenosis);
7. Angiographic thrombus;
8. Target lesion in surgical graft;
9. Total occlusion (TIMI anterograde flow 0 or 1);
10. Ostial lesion;
11. The target lesion bifurcation with side branch that may require intervention during the procedure, with or without stenting;
12. Injuries that are impossible to anticipate predilatation successfully or that is necessary to use rotablator;
13. The target vessel with excessive tortuosity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Lumen Loss | 9 months after the procedure
  For an accurate assessment of the stent conditions 9 months after implantation, a follow-up catheterization will be performed at the 9 months visit in order to measure the diameter of the artery at the stented site.
  A subgroup of 60 patients will be evaluated with volumetric intravascular ultrasound at 9 months. Also, a subgroup of 21 patients will be evaluated with optical coherence tomography at the end of the index procedure and 9 months.

SECONDARY OUTCOMES:
Adverse Cardiac Events | 30 days, 4, 9, 12 months and 2, 3, 4, 5 years after the procedure.
  The clinical follow-up should be performed during the index procedure at 30 days, 4, 9, 12 months and 2, 3, 4, 5 years after the procedure, and should consist of an assessment of the angina status (according to the Canadian Cardiovascular Society Classification and the Braunwald for unstable angina) and major adverse cardiac avents and any interventional treatment (e.g: repeated targetlesion revascularization or recurrent ischemia)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lemos, Principal Investigator — Instituto do Coração - Incor
Locations (10):
- Brazil (10):
  - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Encore - Cardiologia e Radiologia Intervencionista, Goiânia, Goiás
  - Hospital Cardiologico Costantini, Curitiba, Paraná
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Bandeirantes de São Paulo, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto de Assistência Médica ao Servidor Publico Estadual, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo

REFERENCES:
- [Derived] Lemos PA, Abizaid AA, Meireles GC, Sarmento-Leite R, Prudente M, Cantarelli M, Dourado AD, Mariani J Jr, Perin MA, Costantini C, Costa RA, Costa JR, Chamie D, Campos CA, Ribeiro E. Metallic Limus-Eluting Stents Abluminally Coated with Biodegradable Polymers: Angiographic and Clinical Comparison of a Novel Ultra-Thin Sirolimus Stent Versus Biolimus Stent in the DESTINY Randomized Trial. Cardiovasc Ther. 2015 Dec;33(6):367-71. doi: 10.1111/1755-5922.12159. PMID 26352896
- See also: Sponsor site — http://www.scitechmed.com
- See also: National Information System on Ethics in Research Involving Human — http://portal2.saude.gov.br/sisnep